CLINICAL TRIAL: NCT01049295
Title: The Effects of Omega-3 Fatty Acids on Chemotherapy-induced Neuropathy and Inflammation in Patients With Breast Cancer
Brief Title: Omega-3 Fatty Acids and Chemotherapy-induced Neuropathy and Inflammation in Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zohreh Ghoreishi, Master of Nutrition, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 88-04-27-9683
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer
Keywords: taxanes; breast cancer; n3 fatty acids; inflammation
MeSH Terms: conditions — Breast Neoplasms; Inflammation | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oil fish pearls (Experimental): patients with invasive breast cancer who received 640 mg oil fish pearls 3 times a day
  Interventions: Dietary Supplement: oil fish
- placebo (Placebo Comparator): patient with invasive breast cancer who received corn oil pearls as placebo 3 times a day
  Interventions: Other: corn oil pearls

INTERVENTIONS:
Dietary Supplement: oil fish — Active Comparator:640 mg oral oil fish pearls( 54% DHA, 10% EPA) 3 times a day
  Arms: oil fish pearls
Other: corn oil pearls — corn oil pearls 3 times a day
  Arms: placebo

SUMMARY:
The aim of this study is to assess the effects of n-3 fatty acids on taxane-induced neuropathy and neurotoxic inflammatory agents in patients suffering from invasive breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women. Chemotherapy with taxanes in patients with breast cancer causes some complications and neuropathy is one of the most frequent that is dose limiting and even may cause to stop the therapy. n-3 fatty acids have very significant role in improvement the function of the neurons.n-3 fatty acids decrease the demyelination and toxicities resulting from taxanes. They also lower the level of of the neurotoxic inflammatory agents. So,n-3 fatty acids improve the quality of life in this patients. 52 patients with invasive breast cancer will be randomized in a double-blind placebo-controlled manner to receive either 640 mg oil fish pearls( 54% DHA, 10% EPA) 3 times a day or placebo( corn oil pearls) for 3 months(during the chemotherapy with taxanes). Neuropathy (using EMG-NCV test)and the level of IL-1,IL-6, TNF-alpha, hs-crp and serum level of EPA and DHA fatty acids will be measured before chemotherapy with taxanes and at the end of the therapy (after 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Suffering from invasive breast cancer,not receiving any form of supplementations and oil fish

Exclusion Criteria:

* Suffering from the diseases leading to neuropathy, e.g.diabetes, hyperthyroidism, AIDS and primary neural diseases
* Suffering from any other kind of malignancies
* Receiving any chemotherapeutical agents in the past

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-11 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
The EMG-NCV test,The serum level of IL-1,IL-6,TNF-alpha and hs-CRP | first day and after 3 months (before chemotherapy with taxanes and at the end of the therapy

SECONDARY OUTCOMES:
The serum level of DHA and EPA fatty acids | first day and after 3 months( before chemotherapy with taxanes and at the end of the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Ali Keshavarz, professor, Principal Investigator — Tehran University of Medical Sciences; Zohreh Ghoreishi, Ph.D student, Study Director — Tehran University of Medical Sciences
Locations (1):
- : Tehran University of Medical Sciences, School of Public Health, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Ghoreishi Z, Esfahani A, Djazayeri A, Djalali M, Golestan B, Ayromlou H, Hashemzade S, Asghari Jafarabadi M, Montazeri V, Keshavarz SA, Darabi M. Omega-3 fatty acids are protective against paclitaxel-induced peripheral neuropathy: a randomized double-blind placebo controlled trial. BMC Cancer. 2012 Aug 15;12:355. doi: 10.1186/1471-2407-12-355. PMID 22894640